CLINICAL TRIAL: NCT05905224
Title: A Randomized Clinical Trial to Assess the Efficacy of Reducing the Aligners' Wear Protocol on the Predictability of Orthodontic Tooth Movement
Brief Title: Clinical Trial to Assess the Efficacy of Reducing the Aligners' Wear Protocol
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202300981
Record Dates: First submitted 2023-05-04; First posted 2023-06-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-03

CONDITIONS: Orthodontic Tooth Movement
Keywords: clear aligners; wear protocol; 3-day wear; 7-day wear; rate and amount of tooth movement; accuracy; outcomes
MeSH Terms: interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Control) (Active Comparator)
  Interventions: Device: Invisalign 7-day wear protocol
- Group 2 (Experimental) (Experimental)
  Interventions: Device: Invisalign 3-day wear protocol

INTERVENTIONS:
Device: Invisalign 7-day wear protocol — Clear Aligners' (Invisalign, Align technology, San Jose, Calif) 7-day wear protocol
  Arms: Group 1 (Control)
Device: Invisalign 3-day wear protocol — Clear Aligners' (Invisalign, Align technology, San Jose, Calif) 3-day wear protocol
  Arms: Group 2 (Experimental)

SUMMARY:
The hypothesis of this project is that replacing the current 7-day wear protocol with a 3-day wear protocol, while integrating less tooth movement per aligner (reduce the amount of activation per aligner) may produce more consistent and continues orthodontic forces, therefore, increase the predictability, accuracy and outcomes achieved for various types of tooth movements and enhance the rate of tooth movement with the Invisalign system

DETAILED DESCRIPTION:
This randomized clinical trial aims to assess the effectiveness of increasing the frequency of change per aligner, within the standard of care, on the efficacy of achieving better treatment outcomes. We will study the influence of reducing the wear scheduled for Invisalign clear aligners, from 7-day change per aligner to 3-day change per aligner, on the predictability and accuracy of different orthodontic tooth movements by comparing the simulated predicted final outcomes to those achieved at the end of treatment between the two change protocols.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy with no relevant allergies or medical problems
* Male or female between the age of 18 and 30.
* Full permanent dentition except for the third molars
* Class I crowded dentition primarily for the lower anterior teeth (moderate crowding - 4-6 mm - according to Little's Irregularity Index)
* Good oral hygiene and absence of periodontal disease
* Malocclusion to be treated with Invisalign aligners (SmartTrack)
* Any ethnic group

Exclusion Criteria:

* Orthognathic surgical cases
* An extraction treatment plan
* Poor oral hygiene
* Patients with syndromes or craniofacial anomalies.
* The use of any other orthodontic appliance than clear aligners' (Invisalign)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
predictability of the different orthodontic tooth achieved in each of the studies groups movements achieved at the end of treatment in each of the studied groups (3-day wear vs 7-day wear). | 14 months
  assess the influence of reducing the wear scheduled for Invisalign clear aligners, from 7- day wear to 3-day wear, on the predictability and accuracy of different orthodontic tooth movements by comparing the simulated predicted final outcomes to those achieved at the end of treatment between the two wear protocols.
rate of tooth movement for the lower anterior teeth as detected by the consecutive scans captured by the scan box (Dental Monitoring®) in the first 8 weeks of treatment | 2 months
  compare and quantify the magnitude and rate of orthodontic tooth movement between the suggested (3-day) and conventional (7-day) wear protocols for the Invisalign® system using the Dental Monitoring superimposed scans and the data collected from their online platform in the first 8 weeks after Invisalign delivery.

SECONDARY OUTCOMES:
duration of treatment | 14 months
  the total time needed to complete treatment
number of refinements and visits needed for each wear protocol. | 14 months
  the number of additional mid adjustment treatment scans needed for each included subject during the clinical trial duration
Occlusal outcomes | 14 months
  The Peer Assessment rate and/or ABO grading system will be used to measure the final occlusal outcomes achieved in both groups for them to be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Abu Arqub, DDS, Principal Investigator — University of Florida
Locations (1):
- University of Florida _ Department of Orthodontics, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No